CLINICAL TRIAL: NCT03442933
Title: Assessment of the Acute Effect of Cycling Practice in Lumbar and Thigh Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Gerson Garrosa Martín, Gerson Garrosa Martín, PhD Candidate, Universidad Europea de Madrid
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016/UEM18
Record Dates: First submitted 2017-12-14; First posted 2018-02-22 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Physical Endurance; Muscle Fatigue; Musculoskeletal Pain; Muscle Tightness
Keywords: Muscle Fatigue; Cycling; MTB; Tensiomiography
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: A cross-over study with a single group (n = 40) of amateur cyclists subjected to each 2 different intervention conditions: a road bike time trial (CA) and a mountain bike time trial (MT).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Road Cycling first, then Mountain Biking (Active Comparator): First Intervention (3 hours: Road cycling), followed by a 7 days washout, and the second Intervention (3 hours: Mountain Biking).
  Interventions: Other: 3 hours Road Cycling Time Trial; Other: 3 hours Mountain Biking Time Trial
- Mountain Biking first, then Road Cycling (Active Comparator): First Intervention (3 hours: Mountain Biking), followed by a 7 days washout, and the second Intervention (3 hours: Road cycling).
  Interventions: Other: 3 hours Road Cycling Time Trial; Other: 3 hours Mountain Biking Time Trial

INTERVENTIONS:
Other: 3 hours Road Cycling Time Trial — The road itinerary is a mixed route profile of 90 km, an elevation gain of 900 m, with mixed sections, flat, uphill and down over roads with little traffic.
Other: 3 hours Mountain Biking Time Trial — The mountain itinerary, is a mixed route of 55 km, an elevation gain of 600 m, with sections of wide tracks and trails, flat, uphill and down, with a medium technical difficulty.

SUMMARY:
Introduction: Cycling represents a very important level of practice, being among the most practiced sports in Spain. As in any other sport discipline, its practice is associated with the appearance of overloads and sports injuries. Specifically, the 2 most affected areas are the lumbar and knee areas, with an annual prevalence of 58% and 36%, respectively. There is no clear hypothesis to explain the low back pain associated with the practice of cycling, but several authors agree that it may be due to holding an inverted posture of the rachis and the characteristics associated with this sport: long duration, static posture, high intensities, vibrations generated by the terrain, and so forth. The project proposes to analyze the acute effect of a long-lasting bicycle trip (3 hours) on the muscles involved in low back and knee pain, see, lumbar paravertebral, quadriceps and hamstrings, by means of tensiomyography (TMG).

Objectives: the main objective of this study is to evaluate the behavior of the mechanical characteristics of the lower back and thigh muscles, by means of tensiomyography, in amateur cyclists after an acute effort on road and mountain bikes, and to study their possible relationship with low back pain (LBP).

DETAILED DESCRIPTION:
A crossover randomized controlled trial. The participation in the study requires only 2 assistances to the data takings that will be developed in the training laboratory of the Faculty of Sciences of Physical Activity and Sport of the European University. 40 amateur cyclists will be randomly assigned to carry out each (2) conditions of intervention: a road bike time trial (CA) and a mountain bike time trial (MT) separated by 7 days washout. *Randomization marks the order in which participants are subjected to an intervention condition or other.

These sessions will begin with an initial assessment, which will be carried out: an anthropometric assessment (height and weight), followed to an evaluation of the tensiomyographic variable maximal radial displacement (Dm) over the thigh muscles: vastus medialis (VM), rectus femoris (RF), vastus lateralis (VL), biceps femoris (BF), and erector spinae (EE) at the lumbar level, before and after an acute effort (> 3 hours) in CA and MT bicycle. Respect to pain assessment, it will be measured the intensity pain perception on the lumbar region (LBPP) by using a 0 to 10 numeric pain-rating scale; the pressure pain threshold (PPT) with a manual mechanical algometer; and the functional disability caused by LBP through the Roland-Morris Questionnaire (RMQ).

ELIGIBILITY:
Inclusion Criteria:

* Be a man
* Aged between 18 and 55 years.
* Minimum experience in the practice of cycling over 3 years
* Accumulate at least 200 hours of training each year.
* Not having received specific treatment in the musculature evaluated in the last 4 weeks, or being subjected to any treatment at present.
* No pathology diagnosed in the anatomical regions interested in the study (lumbar, thigh, hip or knee).
* Sign the informed consent.

Exclusion criteria

* Have had strenuous exercise in the previous 48 hours
* Having taken energy drinks in the last 48 hours
* Have ingested alcohol or caffeine in the 3 hours prior to taking data.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 40 participants were randomly assigned to their Arm/Group, in which the intervention was administered in 2 different sequences of intervention: 1) Road Cycling first, then Mountain Biking; and 2) Mountain Biking first, then Road Cycling.
Pre-assignment Details: They were required to attend on 2 different occasions to our installation, both spaced a week apart as washout.
Groups:
- Road Cycling First, Then Mountain Biking: They will be examined before and after 3 hours road cycling time trial (TT). And after 7 days washout, they will be examined before and after 3 hours mountain biking TT.
- Mountain Biking First, Then Road Cycling.: They will be examined before and after 3 hours mountain biking time trial (TT). And after 7 days washout, they will be examined before and after 3 hours road cycling TT.
Period: Overall Study
Arm/Group | Road Cycling First, Then Mountain Biking | Mountain Biking First, Then Road Cycling.
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Amateur males from mixed cycling modalities with an experience in the practice of cycling greater than 3 years.
Groups:
- All Study Participants: Regardless of the Arm/Group in which the participants were initially assigned, all participants received all interventions. Therefore they are represented combined into one single Arm/Group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 40
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 40
Height [Mean (Standard Deviation); unit: cm] | 177 (7)
Weight [Mean (Standard Deviation); unit: kg] | 74.4 (8.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain Perception (LBPP)
Description: This variable records the intensity pain perceived on the lumbar region (LBPP) by using a 0 to 10 numeric pain-rating scale (NPRS). This is an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). The LBPP was measured before and after completing each time trial.
Time Frame: Change between Baseline and 3 hours
Population: Amateur males from mixed cycling modalities with an experience in the practice of cycling greater than 3 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Road Cycling First, Then Mountain Biking | Mountain Biking First, Then Road Cycling
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 1 (1.4) | 0.8 (1.2)
  After 3 hours | 3.4 (2.2) | 3.3 (2)

2. Primary Outcome: Maximal Radial Displacement (Dm)
Description: The variable Dm is given by the radial displacement of the muscular belly in a transverse plane, expressed in milimeters (mm) and depends on muscle tone or stiffness. A low Dm is related to a high muscle tone or an excess of stiffness, while a high Dm value indicates a lack of muscle tone or stiffness defect.
Time Frame: Baseline and after 3 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Road Cycling First, Then Mountain Biking | Mountain Biking First, Then Road Cycling.
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 7.6 (2.1) | 7.2 (2.2)
  After 3 hours | 9 (2.1) | 8.8 (2.3)

3. Primary Outcome: Pressure Pain Threshold (PPT)
Description: Measured from 0 to 10kg/cm2 with a manual mechanical algometer (FDK/FDN, Wagner Instruments, 1217 Greenwich, CT 06836), which has bilaterally shown an excellent reliability, reproducibility, and sensitivity on the lumbar erector spinae muscles.
Time Frame: Baseline and after 3 hours
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Road Cycling First, Then Mountain Biking | Mountain Biking First, Then Road Cycling.
Number analyzed (Participants) | 20 | 20
kg/cm^2
  Baseline | 5 (2) | 4.7 (1.9)
  After 3 hours | 4.6 (1.9) | 4.5 (1.8)

4. Secondary Outcome: Roland-Morris Questionnaire (RMQ)
Description: The functional disability caused by LBP through the Roland-Morris Questionnaire (RMQ). The score ranges from 0 to 24, with 0 indicating no disability and 24 maximum disability.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Participants
  Score of 0 | 22
  Score of 1 | 9
  Score of 2 | 3
  Score of 3 | 2
  Score of 4 | 0
  Score of 5 | 1
  Score of 6 | 3
  Score of more than 6 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed.
Arm/Group | Road Cycling First, Then Mountain Biking | Mountain Biking First, Then Road Cycling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT03442933/Prot_SAP_ICF_000.pdf